CLINICAL TRIAL: NCT02915315
Title: Genetics Study of Salt-Sensitive Hypertension in a Chinese Population
Brief Title: Salt-sensitive Hypertension Study in Lantian County
Acronym: SHSL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: NSFC(81570381)
Record Dates: First submitted 2016-09-21; First posted 2016-09-27 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: blood pressure; Hypertrophy; Left Ventricular; arterial Stiffness; Proteinuria; baPWV; ambulatory Blood Pressure
MeSH Terms: conditions — Hypertension; Hypertrophy; Proteinuria | interventions — Salts; Sodium Chloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lantian county adult salt-sensitive hypertension study is a family-based dietary interventional study. Whole blood specimen was collected from each participant who underwent a chronic salt load and potassium supplementation trial.Genomic DNA was extracted from whole blood specimen using the GOLDMAG Whole Blood Genomic DNA Purification Kit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Baseline survey period: All subjects will continue a normal diet for 3 days in which questionnaire design and anthropometric measurements will be implemented.
- Low-salt diet: All subjects will be instructed to maintain a low-salt diet for 7 days (3g of salt or 51.3mmol of sodium per day).
  Interventions: Dietary Supplement: salt
- High -salt diet: After washout period, all subjects will be instructed to maintain a 18g of salt or 307.8mmol of sodium per day.
  Interventions: Dietary Supplement: salt

INTERVENTIONS:
Dietary Supplement: salt — The protocol comprise a questionnaire survey and physical examination during a 3-day baseline observation period, a low-salt diet for 7 days (3g of salt per day) and a high-salt diet for 7 days (18g of salt per day). During the baseline period, each subject is given detailed dietary instructions to avoid table salt, cooking salt, and high-salt foods for the 17-day study duration. To ensure compliance of study participants with the intervention program, they are required to have their breakfast, lunch, and dinner at the study kitchen under supervision of the study staff during the entire study period. All foods are cooked without salt. Onsite study staff members add repackaged salt to the meals of individual subjects as indicated by the study protocol.
  Other Names: Sodium Chloride
  Groups: High -salt diet; Low-salt diet

SUMMARY:
Essential hypertension is a complex trait which results from interaction between environmental factors and genetic factors. Our study aimed to detect the differential expression of LncRNAs and epigenetic changes such as DNA methylation associated with salt sensitive hypertension in human based on a chronic salt loading study conducted in Lantian county, China. Firstly, a chronic salt loading study will be conducted in a Chinese population to differentiate salt-sensitive and salt-resistant individuals. Second, LncRNAs and DNA methylation Chip analysis will be performed using samples collected from salt-sensitive and salt resistant individual, and the results will be analyzed by modern bioinformatics methods to seek for differential genetic markers. In addition, the investigators also try to examine the effects of chronic salt loading on BP, ambulatory BP, microalbuminuria and baPWV and other biochemical indexes. This project had great significance to reveal molecular genetics mechanism in the development of salt, salt-sensitive and hypertension.

DETAILED DESCRIPTION:
The main contents include: (1) Questionnaire design: questionnaire is designed according to the research contents and purposes. The standard questionnaires will be used to collect the general information, dietary habits, lifestyle, medical history and family history etc.(2)Anthropometric measurements: blood pressure, height, body weight, waist and hip, pulse will be acquired by medical practitioners who received professional trainings based on World Health Organization (WHO) standards, and passed relevant examinations.(3) Dietary intervention: The dietary intervention comprise a 3-day baseline observation period, a low-salt diet for 7 days (3g of salt or 51.3mmol of sodium per day) and a high-salt diet for 7 days (18g of salt or 307.8mmol of sodium per day). During the baseline period, each subject is given detailed dietary instructions to avoid table salt, cooking salt, and high-salt foods for the 21-day study duration. To ensure compliance of study participants with the intervention program, they are required to have their breakfast, lunch, and dinner at the study kitchen under supervision of the study staff during the entire study period. All foods are cooked without salt. Onsite study staff members add prepackaged salt to the meals of individual subjects as indicated by the study protocol. (4) Blood and urine samples collection: morning fasting blood, nocturnal enuresis, and 24-hour urine specimen will be collected by medical staffs, and blind tubes will be set up according to 5% of the total samples. Blood biochemistries including serum total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, fasting glucose, creatinine and hsCRP can be measured using automatic biochemical analyzer. The sodium and potassium concentrations in the urine will be measured by flame photometry. The total sodium and potassium excretions in urine in 24h were calculated by multiplying the concentration and 24-h volume of urine. (5) DNA methylation and LncRNA detection: Using a method of modifying a hydrogen sulfite salt and gene chip technology to detect DNA methylation and LncRNA. (6) LncRNA: LncRNA will be measured with gene chip technology after the high salt intervention period. (7) Auxiliary examinations: Auxiliary examinations including carotid intima-media thickness, endothelium-dependent vasodilation (FMD), measurements of brachial-ankle pulse wave velocity (baPWV) and electrocardiographic parameters. The measurement will be done in hospitals by medical practitioners who received professional trainings and passed relevant examinations. (8) Data processing and statistics: the investigators should input the data to the database, and utilize software such as SPSS, STATA, Haploview and FBAT to analyze. (9)Quality control: ① Questionnaire is strictly designed and amended by epidemiologist and clinical experts. ② A standardized "Investigator Handbook" will be stipulated according to the guidelines. ③ Staff members are required to do a rigorous training and pass the exam. ④ The investigation process will be strictly supervised by the principal investigator. ⑤ Data entry use the parallel double entry method. ⑥ During laboratory testing, blank control and blind detection are applied to ensure the quality. ⑦Data analysis is performed by 2-3 postgraduates, inconsistent data need to be double checked.

ELIGIBILITY:
Inclusion Criteria:

* Han individuals in rural northern China
* adults aged 18-65 years
* individuals who had a mean systolic BP (SBP) between 130-160 mmHg and/or a diastolic BP (DBP) between 85-100 mmHg and no use of antihypertensive medications were identified as the proband
* the probands'parents,siblings, spouses, and offspring were recruited for the study.

Exclusion Criteria:

* Secondary hypertension
* a history of severe cardiovascular disease
* chronic kidney disease or liver disease
* unable to complete the examination
* unable/refuse to sign the informed consent form

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is ready to recruit from Shaanxi Lantian County, aged 18-65 years old and sex is not limited. The exclusion criteria were hypertension, use of antihypertensive medication, clinical cardiovascular disease, chronic liver disease, chronic kidney disease, or diabetes mellitus, pregnancy, or high alcohol consumption.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-02-28 (Estimated); Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
blood pressure value(mmHg) | The first day of the three-day baseline survey period.
  The study will last approximately 3 months (Oct 2016 to Dec 2016). During this period, each subject will receive a three-day baseline survey examination. Three BPs (mmHg) measurement will be obtained using a Blood Pressure Monitor on the first day of the three-day baseline survey period.

SECONDARY OUTCOMES:
Ambulatory Blood Pressure Monitoring（mmHg） | Second day of the three-day baseline survey period
  The study will last approximately 3 months (Oct 2016 to Dec 2016). During this period, each subject will receive a three-day baseline survey examination. Ambulatory blood pressure（mmHg）will be measured with Omron Ambulatory Blood Pressure Monitor during the three-day baseline survey period
Microalbuminuria（mg/24h） | Second day of the three-day baseline survey period
  The study will last approximately 3 months (Oct 2016 to Dec 2016). During this period, each subject will receive a three-day baseline survey examination. On the second day, 24-hour urinary will be collected and the concentrations of microalbuminuria in the urine sample will be measured with Hitachi biochemical analyzer. The 24-h microalbuminuria（mg/24h）of each subject is calculated as the concentration of microalbuminuria multiplied by the 24-h urine volume of each individual.
Increased arterial stiffness（baPWV,mm/s） | Second day of the three-day baseline survey period
  The study will last approximately 3 months (Oct 2016 to Dec 2016). During this period, each subject will receive a three-day baseline survey examination. Brachial-ankle pulse wave velocity（baPWV, mm/s）will be measured with Noninvasive automatic waveform analyzer during the three-day baseline survey period.
DNA methylation | Last day of the low salt or high salt intervention period
  The study will last approximately 3 months (Oct 2016 to Dec 2016). During this period, each subject will receive a seven-day high salt intervention subsequent to a seven-day low salt intervention. DNA methylation will be measured with a method of modifying a hydrogen sulfite salt at the last day of the low salt or high salt intervention.
LncRNA | Last day of the low salt or high salt intervention period
  The study will last approximately 3 months (Oct 2016 to Dec 2016). During this period, each subject will receive a seven-day high salt intervention subsequent to a seven-day low salt intervention. IncRNA will be measured with gene chip technology at the last day of the low salt or high salt intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Mu, doctor, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mu J, Zheng S, Lian Q, Liu F, Liu Z. Evolution of blood pressure from adolescents to youth in salt sensitivies: a 18-year follow-up study in Hanzhong children cohort. Nutr J. 2012 Sep 14;11:70. doi: 10.1186/1475-2891-11-70. PMID 22978814
- [Result] Liu F, Zheng S, Mu J, Chu C, Wang L, Wang Y, Xiao H, Wang D, Cao Y, Ren K, Liu E, Yuan Z. Common variation in with no-lysine kinase 1 (WNK1) and blood pressure responses to dietary sodium or potassium interventions- family-based association study. Circ J. 2013;77(1):169-74. doi: 10.1253/circj.cj-12-0900. Epub 2012 Oct 12. PMID 23059770
- [Result] Wang Y, Liu FQ, Wang D, Mu JJ, Ren KY, Guo TS, Chu C, Wang L, Geng LK, Yuan ZY. Effect of salt intake and potassium supplementation on serum renalase levels in Chinese adults: a randomized trial. Medicine (Baltimore). 2014 Jul;93(6):e44. doi: 10.1097/MD.0000000000000044. PMID 25058146
- [Derived] Wang Y, Jia H, Gao WH, Zou T, Yao S, Du MF, Zhang XY, Chu C, Liao YY, Chen C, Wang D, Ma Q, Hu JW, Wang KK, Yan Y, Sun Y, Hu GL, Niu ZJ, Zhou HW, Zhang X, Wang X, Li CH, Chen FY, Gao K, Zhang J, Guan YJ, Chang J, Yang TL, Mu JJ. Associations of plasma PAPP-A2 and genetic variations with salt sensitivity, blood pressure changes and hypertension incidence in Chinese adults. J Hypertens. 2021 Sep 1;39(9):1817-1825. doi: 10.1097/HJH.0000000000002846. PMID 33783375
- [Derived] Zhang J, Yin Y, Chen L, Chu C, Wang Y, Lv Y, He M, Martin M, Huang PH, Mu JJ, Shyy JY, Yuan ZY. Short-Term High-Salt Diet Increases Corin Level to Regulate the Salt-Water Balance in Humans and Rodents. Am J Hypertens. 2018 Jan 12;31(2):253-260. doi: 10.1093/ajh/hpx148. PMID 28985241